CLINICAL TRIAL: NCT04553991
Title: Analgesic Effect of Ultrasound-Guided Bilateral Quadratus Lumborum Block (Lateral Approach) Versus Bilateral Transversus Abdominis Plane Block With General Anesthesia in Laparoscopic Abdominal Surgery (Randomized Controlled Clinical Trial)
Brief Title: Lateral Quadratus Lumborum Block Versus Transversus Abdominis Plane Block in Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Mohammed abdelaleem, The Analgesic Effect of Ultrasound-Guided Bilateral Quadratus Lumborum Block (lateral Approach) Versus Bilateral Transversus Abdominis Plane Block with General Anesthesia in Laparoscopic abdominal surgery (Randomized Controlled Clinical Trial), Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: M421
Record Dates: First submitted 2020-09-05; First posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Abdominal Pain
Keywords: laparoscopy; QL block; TAP block
MeSH Terms: conditions — Abdominal Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QL block group (Active Comparator): For the ultrasound-guided quadratus lumborum block group, the patient was placed in lateral position . QL was identified medial to the aponeurosis of transversus abdominis muscle. Then the needle was inserted from supero-anterior to postero-inferior and advanced using in plane technique till the needle tip reached the anterolateral border of the QL at its junction with transversalis fascia.An injection of 20 mL of 0.25% bupivacaine was applied bilaterally
  Interventions: Procedure: Ultrasound guided QL block
- TAP block group (Active Comparator): For the ultrasound-guided TAP block,The probe was placed in the mid-axillary line above the level of the anterior superior iliac spine, then slided cranially till the three abdominal wall muscles identified (External oblique muscle (EAO), internal oblique muscle (IOM) and transverse abdominis muscle (TAM)). The needle was advanced using in-plane technique till it reached the transvers abdominis plane. An injection of 20 mL of 0.25% bupivacaine was applied bilaterally
  Interventions: Procedure: Ultrasound guided TAP block

INTERVENTIONS:
Procedure: Ultrasound guided QL block — 20 mL of 0.25% bupivacaine was applied bilaterally at the anterolateral border of the QL at its junction with transversalis fascia
  Arms: QL block group
Procedure: Ultrasound guided TAP block — 20 mL of 0.25% bupivacaine was applied bilaterally in the TAP
  Arms: TAP block group

SUMMARY:
The transversus abdominis plane (TAP) block is an already established technique and is considered now as an efficient part of the multimodal pain management approach for abdominal surgical procedures. The quadratus lumborum block (QLB) is a recently described regional block that was first described by Blanco et al , which has been reported to provide an effective analgesia for upper and lower abdominal surgeries. The aim of this study is to compare the analgesic efficacy of TAP block and QLB 1 after laparoscopic abdominal surgery regarding opioid consumption, duration of analgesia and visual analog score.

This prospective randomized controlled observer-blinded study compared between the analgesic efficacy between TAP block (n=25) versus QL block (n=25) in patients aged (18-60) years of American society of anesthesiologists physical status class I & II scheduled for elective laparoscopic abdominal surgical procedures. The primary outcome was the cumulative morphine consumption at first 24 hours postoperatively. Secondary outcomes included VAS scores, first analgesic requirements and any postoperative complications

DETAILED DESCRIPTION:
This prospective randomized, observer-blinded paralleled groups study was conducted following the tents of the Declaration of Helsinki. This study was approved by the local institutional ethics committee and local institutional review board of Fayoum university hospital and written informed consent was obtained from 50 adult patients scheduled for elective laparoscopic abdominal surgical procedures (inguinal hernia repair-missed IUCD extraction-appendectomy-ovarian vein ligation) between July 2019 and February 2020.

Patients were randomly allocated into two groups (QLB group n=25 and TAPB group n=25) using computer generated random numbers kept in separate opaque envelopes that were opened by the study investigator just before the block. The patient and the data collector were unaware of the group allocation till the end of the study.

Pre-operative assessment (History, examination and investigations) was done (according to the local protocol designed to evaluate the patients). Demographic characteristics: age, weight, height and BMI were recorded in preoperative assessment of patients. All patients received 150 mg Ranitidine oral tablet at night and on the morning just before the operation as a premedication. Before surgery, the participants received education about the VAS pain score (0-10) (where 0 = no pain and 10 = worst comprehensible pain) and the details of the nerve block procedures. After a 6 hrs fasting, the patients were taken to the operation theatre.

Upon arrival to the operating room standard monitors (Pulse oximeter, noninvasive blood pressure monitoring, capnography and electrocardiogram) were applied and continued all over the operation, an 18 gauge peripheral intravenous (IV) cannula was inserted, IV midazolam 0.03 mgkg-1, metoclopramide 10 mg, and ceftriaxone 1 gm were administered to all patients as premedication then pre-oxygenation with O2 100% for at least 3 min then induction of anesthesia was done with fentanyl 1μgkg-1, propofol 1.5-2 mgkg-1 and atracurium 0.5 mgkg-1. Anesthesia was maintained by volume controlled ventilation (VCV) tidal volume 6-8 mlkg-1 with oxygen and air (50:50) with target of EtCO2≈ 35-40 mmHg, isoflurane 1:1.5 % volume concentration and atracurium 0.1 mgkg-1 every 20-30 minutes.

The study solution was prepared in two syringes each contained 20 ml of bupivacaine 0.25%. By the end of surgery and before recovery from general anesthesia, either blocks were done using a high-frequency ultrasound probe Active Array L12-4 (8-13MHz) of an ultrasound machine (Philips clear vue350, Philips healthcare, Andover MA01810, USA) and a 22-gauge, 50 mm echogenic needle (Stimuplex D; B Braun, Germany).

For the ultrasound-guided quadratus lumborum block group, the patient was placed in lateral position and skin sterilization was done with povidone iodine. Then a high frequency linear probe was placed above the iliac crest to recognize the three layers of the abdominal wall muscles. Transversus abdominis was traced posteriorly until the transversus aponeurosis appeared, then the probe tilted slightly caudal to enhance the appearance of transversus aponeurosis. QL was identified medial to the aponeurosis of transversus abdominis muscle. Then the needle was inserted from supero-anterior to postero-inferior and advanced using in plane technique till the needle tip reached the anterolateral border of the QL at its junction with transversalis fascia. After negative aspiration (to exclude intravascular injection), the correct needle position was confirmed by hydrodissection using 1mL of normal saline. Then 20 mL of 0.25% bupivacaine was applied. The same technique was performed on the other side.

For the ultrasound-guided TAP block, skin sterilization was done with povidone iodine. The probe was placed in the mid-axillary line above the level of the anterior superior iliac spine, then slided cranially till the three abdominal wall muscles identified (External oblique muscle (EAO), internal oblique muscle (IOM) and transverse abdominis muscle (TAM)). The needle was advanced using in-plane technique till it reached the transvers abdominis plane between the IOM and TAM, the correct needle position was proved by hydrodissection using 1 mL of normal saline. An injection of 20 mL of 0.25% bupivacaine was applied. The same technique was performed on the other side.

After performing the block anesthesia was discontinued and tracheal extubation was done once the patient fulfilled the extubation criteria. Patients were transferred to post-anesthetic care unit (PACU), where they were discharged from the PACU after a modified Aldrete score≥9. Visual analogue scale (VAS) was used to assess postoperative pain. All patients received analgesics according to the local institutional protocol as following (paracetamol 1gm IV infusion/8 hrs and ketorolac 30 mg IM/12 hrs.). A postoperative rescue analgesia with morphine sulfate IV was given to patients with VAS >4 at a bolus dose of 3 mg increments with a maximum dose of 15mg per 4 hours or 45mg per 24 hours.

Sample size was estimated using G*Power© software version 3.1.9.2 (Institute of experimental psychology, Heinrich Heine University, Dusseldorf, Germany)149 with total opioid consumption among the two groups as the main primary outcome. Previous similar researches150 demonstrated that the effect size between the two groups was expected to be large of 1.12 and it calculated that 42 patients (21 patients per group) would provide to achieve a power of 95% with type I error rate of 0.05. However, we assigned 50 patients (25 patients per group) to compensate for data loss. The collected data were organized, tabulated and statistically analyzed using SPSS software statistical computer package version 22 (SPSS Inc, USA). Data were tested for normality using shapiro-wilks test. Numerical variables such as age, body weight, height and BMI were normally distributed and were described as mean ± standard deviation (SD). An independent t-test was used to compare the mean values of the two groups. Other variables were not normally distributed and were presented as median and interquartile range (IQR); Mann-Whitney U test was used as a test of significance. The time-to-event variable (time to analgesic request) was evaluated using the Kaplan-Meier method, and the logrank test was used to compare the groups. Qualitative data were presented as numbers and percentages, and the chi-squared test was used to determine significance. A two-sided P-value of <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective laparoscopic abdominal surgeries (inguinal hernia repair-missed IUCD extraction-appendectomy-ovarian vein ligation)
* Patient aged 18-60 years
* American Society of Anesthesiologists Physical Status I or II.

Exclusion Criteria:

* Patient refusal
* Body mass index (BMI) > 40 kilogram/square meter
* Contraindication to regional anesthesia (coagulopathy, allergy to local anesthetic, sever thrombocytopenia or infection at puncture site)
* Sepsis
* Chronic pain condition requiring the intake of opioids at home
* Any significant neurological, cardiovascular or respiratory disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
The total morphine consumption at first 24 hours postoperatively | 24 hours postoperatively
  amount of morphine used in milligram after each block

SECONDARY OUTCOMES:
Postoperative pain, assessed using visual analog scale (VAS) score at 30 min postoperatively. | 30 minutes postoperatively
  from 0 to 10 degrees
Postoperative pain, assessed using visual analog scale (VAS) score at 2 h postoperatively. | 2 hours postoperatively
  from 0 to 10 degrees
Postoperative pain, assessed using visual analog scale (VAS) score at 4 h postoperatively. | 4 hours postoperatively
  from 0 to 10 degrees
Postoperative pain, assessed using visual analog scale (VAS) score at 6 h postoperatively. | 6 hours postoperatively
  from 0 to 10 degrees
Postoperative pain, assessed using visual analog scale (VAS) score at 12 h postoperatively. | 12 hours postoperatively
  from 0 to 10 degrees
Postoperative pain, assessed using visual analog scale (VAS) score at 24 h postoperatively. | 24 hours postoperatively
  from 0 to 10 degrees
Time to the first analgesic request | 24 hours postoperatively
  defined as the time interval elapsed between recovery and the first dose of morphine given.
frequency of patients required postoperative opioid. | First 24 hours postoperatively
  in numbers
incidence of postoperative nausea and vomiting | First 24 hours postoperatively
  Any postoperative nausea or vomiting related to morphine consumption
incidence of postoperative pruritus | First 24 hours postoperatively
  Any postoperative pruritus related to morphine consumption
incidence of postoperative sedation at 30 min postoperatively | at 30 minutes postoperatively
  sedation was assessed with a five-point sedation scale
incidence of postoperative sedation at 2 h postoperatively | at 2 hours postoperatively
  sedation was assessed with a five-point sedation scale
incidence of postoperative sedation at 6 h postoperatively | at 6 hours postoperatively
  sedation was assessed with a five-point sedation scale
incidence of postoperative sedation at 12 h postoperatively | at 12 hours postoperatively
  sedation was assessed with a five-point sedation scale
incidence of postoperative sedation at 24 h postoperatively | at 24 hours postoperatively
  sedation was assessed with a five-point sedation scale
incidence of local anesthetic systemic toxicity | in the first 24 hours postoperatively
  any observed local anesthetic systemic toxicity manifestations including CNS or CVS manifestations
incidence of vascular injury | in the first 24 hours postoperatively
  incidence of vascular injury after each block
incidence of local hematoma | in the first 24 hours postoperatively
  incidence of local hematoma at injection site after each block
incidence of visceral injury | in the first 24 hours postoperatively
  incidence of visceral injury after each block

OTHER OUTCOMES:
Patient's age | 15 minutes before operation
  In years
Patient's weight | 15 minutes before operation
  In kilograms
Patient's height | 15 minutes before operation
  In meters
Body mass index | 15 minutes before operation
  In kilogram/ square meter

CONTACTS AND LOCATIONS:
Overall Officials: Maged L boules, MD, Study Chair — Faculty of medicine, Fayoum university
Locations (1):
- Fayoum University hospital, El Fayoum Qesm, Fayoum Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kumar GD, Gnanasekar N, Kurhekar P, Prasad TK. A Comparative Study of Transversus Abdominis Plane Block versus Quadratus Lumborum Block for Postoperative Analgesia following Lower Abdominal Surgeries: A Prospective Double-blinded Study. Anesth Essays Res. 2018 Oct-Dec;12(4):919-923. doi: 10.4103/aer.AER_158_18. PMID 30662131
- [Background] Okmen K, Metin Okmen B, Topal S. Ultrasound-guided posterior quadratus lumborum block for postoperative pain after laparoscopic cholecystectomy: A randomized controlled double blind study. J Clin Anesth. 2018 Sep;49:112-117. doi: 10.1016/j.jclinane.2018.06.027. Epub 2018 Jun 18. PMID 29929169
- [Derived] Fargaly OS, Boules ML, Hamed MA, Aleem Abbas MA, Shawky MA. Lateral Quadratus Lumborum Block versus Transversus Abdominis Plane Block in Laparoscopic Surgery: A Randomized Controlled Study. Anesthesiol Res Pract. 2022 Mar 28;2022:9201795. doi: 10.1155/2022/9201795. eCollection 2022. PMID 35386840